CLINICAL TRIAL: NCT04880265
Title: Assessing the Burden of Perioperative Atrial Fibrillation in Patients Undergoing Cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jakob Wollborn, MD, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2021P000356
Record Dates: First submitted 2021-04-06; First posted 2021-05-10 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation; Cardiac Surgery
Keywords: Wearable Device
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing cardiac surgery
  Interventions: Device: Vivalink wearable life sensors

INTERVENTIONS:
Device: Vivalink wearable life sensors — Collection of EKG data

SUMMARY:
Background and Significance:

In the United States approximately 220,000 patients undergo cardiac surgery per annum. Among potential complications, the incidence of atrial fibrillation (AF) is estimated at 30 - 60 %, and therefore presents the most common adverse event after cardiac surgery. Multiple complications may be associated with AF: Patients are usually subject to an increased length-of-stay in the intensive care unit and in the hospital. Furthermore, the risk for stroke and development of long-term AF is elevated, while further anticoagulation is required putting the patient at risk for bleeding. On average, an additional $10,000 - $20,000 is spent for each patient with AF. However, the exact burden of postoperative AF still remains unknown.

Specific Aims of Research Project:

1. To collect data from an electrocardiogram (EKG) monitoring patch, we aim to accurately determine the prevalence of atrial fibrillation in patients undergoing cardiac surgery at our center.
2. To collect data on epidemiological characteristics to investigate risk factors for developing perioperative atrial fibrillation in patients undergoing cardiac surgery. This will allow us to create robust risk prediction models.

ELIGIBILITY:
Inclusion Criteria:

* Elective open heart surgery
* Age > 20 years

Exclusion Criteria:

* Refusal to participate (patient or health care proxy)
* Participation in other pharmacological trials
* Lack of data or poor data quality which cannot be analyzed for any heart rhythm in 80% of the postoperative study period.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing cardiac surgery
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Atrial Fibrillation | Up to 30 days after discharge from the hospital
  Atrial Fibrillation

SECONDARY OUTCOMES:
Other arrhythmias | Up to 30 days after discharge from the hospital
  Other arrhythmias

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States